CLINICAL TRIAL: NCT05964127
Title: Local and Systemic Effects of Peri-implantitis and Its Treatment (LASSO). A Randomised Controlled Clinical Trial
Brief Title: Peri-implantitis and Systemic Inflammation
Acronym: LASSO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eastman Dental Insitute and Hospital (Other)
Responsible Party: Principal Investigator, Prof Francesco D'Aiuto, Professor & Head of Department of Periodontology, Eastman Dental Insitute and Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EDGE ID 124712
Record Dates: First submitted 2020-12-11; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Peri-Implantitis and Systemic Inflammation
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A - Non-surgical hand instruments (Active Comparator): After appropriate local anaesthesia of the treatment site supragingival, subgingival and implant surface debridement will be undertaken with Hu-Friedy titanium implant hand instruments only. Any remaining supragingival deposits will be polished using a contra-angle handpiece, rubber cup and Cleanic polishing paste.
  Interventions: Other: Hand instruments
- Group B - Non-surgical Air-flow (Active Comparator): After appropriate local anaesthesia of the treatment site supragingival, subgingival and implant surface debridement will be undertaken using EMS PerioFlow with Plus powder (Erythritol) and supplemented with EMS Piezon and EMS AirFlow and Plus powder as required.
  Interventions: Device: Air flow device
- Group C - Surgical Air-flow (Active Comparator): After appropriate local anaesthesia of the treatment site a full thickness mucoperiosteal flap will be raised to adequately expose the tissue defect. Supragingival, subgingival and implant surface debridement will be undertaken using EMS PerioFlow with Plus powder (Erythritol) and supplemented with EMS Piezon and EMS AirFlow and Plus powder as required.
  Interventions: Device: Air flow device; Procedure: Access flap surgery

INTERVENTIONS:
Device: Air flow device — An air/powder device for surface decontamination
  Arms: Group B - Non-surgical Air-flow; Group C - Surgical Air-flow
Other: Hand instruments — Periodontal hand instruments
  Arms: Group A - Non-surgical hand instruments
Procedure: Access flap surgery — To improve the surgical access for implant decontamination
  Arms: Group C - Surgical Air-flow

SUMMARY:
To investigate the effects of peri-implantitis (a disease around dental implants) and its treatment at both local and systemic levels using clinical and biological parameters.

One study with two parts which will run simultaneously. An initial observational study comparing cases and controls and a subsequent interventional study in which the cases will proceed to treatments and all participants will be followed up for 6 months.

DETAILED DESCRIPTION:
Dental implants provide the gold standard treatment modality for missing teeth in most clinical situations. However, patient-related, site-related and clinician-related factors play a significant part in the management of patents with edentulous spaces. As the provision of implants increases worldwide and as patient life expectancy increases the long-term maintenance of implants and their restorative components will be essential. Similar to periodontal disease occurring in the periodontium around teeth there is an akin peri-implant disease process occurring in the peri-implant mucosa around implants. The prevalence of peri-implantitis in studies range from 1-47%, with an estimated weighted mean prevalence of 22%. Systematic analysis at implant-based and subjected-based levels shows prevalence's of peri-implantitis of 9.25% and 19.83% respectively.

Peri-implantitis is an inflammatory disease of the soft tissues around an osseointegrated dental implant accompanied by bone loss beyond normal physiological remodelling. Like periodontitis, peri-implantitis is the result of a host inflammatory response to a microbial biofilm, which results in inflammation of the peri-implant connective tissue and progressive bone loss. The current understanding, although limited, suggests that peri-implant disease is a condition that, whilst having several traits in common with periodontal disease, is unique, with distinctive features. Recent discoveries in microbiology opens a completely new perspective on the aetiology of peri-implant disease and the further development of metagenomics might open the way to new therapeutic approaches.

Systemic inflammation plays a crucial role in a number of chronic disorders including diabetes and cardiovascular diseases. There is consistent and substantial evidence proposing that inflammation plays a causative role in the onset and progression of these chronic disorders. Periodontitis is linked to systemic inflammation and effective periodontal treatment resolves this host response. It is plausible to suggest that peri-implantitis could well represent a similar inflammatory trigger for the host. Recent experimental human evidence has confirmed peri-implantitis is associated with a larger mucosal inflammatory infiltrate. This local mucosal response and possible bacterial dissemination, could be triggering a systemic inflammatory response, as assessed by elevated levels of a common inflammatory biomarkers, called C-reactive protein (CRP).

With an inflammatory pathophysiology an exploration of key inflammatory biomarkers can help in disease quantification. Whilst peri-implant crevicular fluid (PICF) will be an area to assess for inflammatory biomarkers of peri-implantitis the focus is still on the blood-borne systemic inflammatory challenge, specifically focusing on the acute-phase protein CRP. CRP is a pentameric pattern recognition molecule which is extremely sensitive to the systemic response to inflammation and regulated by key cytokines like Interleukin 6 (IL-6).

Evidence on CRP specifically within peri-implant disease is lacking. However, studies which use CRP to assist in the diagnosis of diseases around other implantable biomaterials i.e. prosthetic hip and knee joint infections are available and show benefits when combined with other diagnostic tests. Increased levels of CRP have been observed in gingivitis and periodontitis reflecting the locally stressed environment. However, CRP levels fluctuate with various confounding factors including aging, elevated triglycerides and insulin-resistance diabetes. Clinical trials have also shown that treatment for periodontal infection with intensive mechanical therapy can significantly lower the serum CRP levels.

Currently the management of peri-implantitis is somewhat variable and relies on our knowledge and understanding of the management of periodontitis. The need for implant surface decontamination is unequivocal, however, the implant surface is incomparable to that of a tooth root surface. Treatment options include, and often combine, non-surgical mechanical instrumentation, with or without adjunctive antimicrobials, to surgeries ranging from simple access flaps for open flap debridement, with or without osseous recontouring, to implantoplasty and defect regeneration using biomaterials. Systematic reviews have attempted to collate the evidence to provide some management clarity but fell short due to the variability in peri-implantitis case definitions and high heterogeneity of included studies. The challenges of successful instrumentation of implants is that the macro-topography has voids which are smaller than the width of the narrowest surgical instruments. A novel approach to this conundrum is the decontamination of the implant surface using an air-powder abrasive system. Such a technique has been shown, under in vitro evaluation, to remove 99.9% of bacteria from the test specimens.

Peri-implantitis treatment is not currently as predictable as for periodontitis and there must be a focus for innovative treatment approaches. We have strong evidence to support the expected clinical outcomes of non-surgical periodontal therapy and access flap periodontal surgery in periodontitis. The equivalent evidence in peri-implantitis treatment is lacking, in part, due to the challenges of decontamination of an implant surface. The use of air-powder abrasion systems may be an area worthy of further research to determine if this technically appropriate treatment provides clinical evidence of success through appropriately designed trials. The EMS designed PerioFlow system is such a system which combines air-powder-water delivered through a multi-outlet, flexible, single-use nozzle.

This study is therefore aimed at assessing the potential effects of peri-implantitis and different treatment approaches on both peri-implant inflammation and systemic inflammation. The study is conceived into two parts. One part investigating the association between peri-implantitis and local and systemic inflammation as measured through systemic inflammatory biomarkers, like CRP, in saliva, PICF and blood, but additionally reporting on any differences in the clinical parameters, microbiology, soft tissue thickness and vascularity between health and peri-implantitis. The second part focuses on three different treatment modalities for peri-implantitis and compares the outcomes of these using the same clinical, microbiological, immunological and vascular parameters.

This study will allow us to identify any associations, quantify the effects, postulate the potential clinical implications, evaluate clinical treatments and guide future interventional studies.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age and in good general health
* A minimum of 20 teeth
* Participants must have at least one implant in situ with peri-implantitis as per its case definition
* Must voluntarily agree to sign the consent form

Exclusion Criteria:

* Currently on any weight reduction program
* History of diabetes
* Uncontrolled or currently undergoing treatment for systemic medical conditions
* Chronic treatment (defined as 2 weeks or more) of antibiotic, anti-inflammatory or anticoagulant therapy during the month preceding the baseline assessment
* Taking statins drugs
* History of alcohol or drug abuse
* Self-reported pregnancy or breastfeeding
* Patients who have active periodontitis as per its case definition and/or have had treatment for periodontitis within the last 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Inflammation | 6-months after treatment
  Serum CRP

SECONDARY OUTCOMES:
Inflammation | Baseline, 3 and 6-months after treatment
  IL-6
Endothelial Function | Baseline, 3 and 6 months after treatment
  FMD
OCT | Baseline, 3 and 6 months after treatment
  Gingival epithelial inflammatory status using Optical Coherence Tomography (OCT)
Blood flow | Baseline, 3 and 6 months
  Gingival vascularity using Laser Speckle Contrast Imager (LSCI)
Gingival tissue thickness | Baseline, 3 and 6 months after treatment
  Ultrasound gingival assessment

CONTACTS AND LOCATIONS:
Locations (1):
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided